CLINICAL TRIAL: NCT03881709
Title: The Efficacy of Decision Support E-book for Reducing Decisional Conflict on Prostate Biopsy Decision Making in Patients With Elevated Prostate-specific Antigen
Brief Title: The Efficacy of Decision Support E-book for Prostate Biopsy Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: (667)107A-39
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Prostate-Specific Antigen
Keywords: prostate biopsy; E-Book; decision support intervention; decision self-efficacy; decision conflict

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group will receive the biopsy decision support intervention delivered by a nurse using an E-Book containing a comprehensive information about prostate biopsy.
  Interventions: Behavioral: Using an E-Book
- The control group (No Intervention): The control group will receive a health education about prostate biopsy.

INTERVENTIONS:
Behavioral: Using an E-Book — The intervention group will receive the biopsy decision support intervention delivered by a nurse using an E-Book containing a comprehensive information about prostate biopsy.
  Arms: The intervention group

SUMMARY:
PURPOSE: This study is to test the efficacy of decision support E-Book for 1) increasing prostate biopsy knowledge and decision self-efficacy, and 2) reducing decisional conflict on prostate biopsy decision making in patients with elevated serum PSA.

DESIGN: The study is based on an experimental design. A convent sample of 110 adult males with a PSA greater than 4.0 ng/mL and the transrectal ultrasound-guided prostate biopsy suggested by a physician will be recruited from the urology clinics. Patients will be randomly assigned to the intervention and control group. The intervention group will receive the biopsy decision support intervention delivered by a nurse using an E-Book containing a comprehensive information about prostate biopsy. The control group will receive a health education about prostate biopsy. Data on biopsy knowledge, decision self-efficacy and decision conflict will be collected at pre and post test by using the study questionnaires.

ANALYSIS: Independent sample t -tests and chi-square tests will be used to compare the between group baseline equilibrium. Independent sample t -tests will be also used to analyze the between group differences in biopsy knowledge, decision self-efficacy, and decision conflict at post-test to evaluate the efficacy of the decision support intervention.

DETAILED DESCRIPTION:
Prostate-specific antigen (PSA) is the primary screening test for prostate cancer. The elevated PSA test result is usually followed by the transrectal ultrasound-guided prostate biopsy (TRUS-Bx) for further diagnosis. However, patients often have lots concerns while deciding whether or not to undergo a prostate biopsy. They may worry about the biopsy associated complications such as urinary tract infection, pain, hematuria, bloody stools, etc., causing damage to urinary tract or sexual function, diagnosed with prostate cancer, or cancer spreading. Some may even worry about that a cancer cell can be transmitted to a partner through sexual activity after a biopsy. All these can cause physiological stress and decisional conflict for the patients. Therefore, it is necessary to provide decision support measures in order to improve the patients' knowledge regarding the advantages and disadvantages of prostate biopsy, to increase their decision self-efficacy, and to decrease their decisional conflict, thereby to achieve the share decision making goal. However, few studies have examined the efficacy of decision aids on prostate biopsy decision making. Therefore, the purpose of this study is to test the efficacy of decision support E-Book for 1) increasing prostate biopsy knowledge and decision self-efficacy, and 2) reducing decisional conflict on prostate biopsy decision making in patients with elevated serum PSA.

The study is based on an experimental design. A convent sample of 110 adult males with a PSA greater than 4.0 ng/mL and the transrectal ultrasound-guided prostate biopsy suggested by a physician will be recruited from the urology clinics. Patients will be randomly assigned to the intervention and control group. The intervention group will receive the biopsy decision support intervention delivered by a nurse using an E-Book containing a comprehensive information about prostate biopsy. The control group will receive a health education about prostate biopsy. Data on biopsy knowledge, decision self-efficacy and decision conflict will be collected at pre and post test by using the study questionnaires. The study instruments include the prostate biopsy knowledge scale, the Decision Self-Efficacy Scale, and the Decisional Conflict Scale. Data on whether the patients received a prostate biopsy will also be collected from the patients' medical records.

Independent sample t -tests and chi-square tests will be used to compare the between group baseline equilibrium. Independent sample t -tests will be also used to analyze the between group differences in biopsy knowledge, decision self-efficacy, and decision conflict at post-test to evaluate the efficacy of the decision support intervention.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 40-80
2. PSA greater than 4.0 ng/mL
3. the transrectal ultrasound-guided prostate biopsy suggested by a physician
4. able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

1. had been diagnosed with prostate cancer
2. had been diagnosed with psychiatric diseases
3. with cognition impairments

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Prostate Biopsy Knowledge Scale | 1 hour after pre-test
  The scale measures patient's knowledge of prostate biopsy. There are 16 items in the scale. Each item is rated on dichotomy. The possible score for the scale ranges from 0 to 16. The higher values represent more knowledge of prostate biopsy patient have.
Decision Self-Efficacy Scale | 1 hour after pre-test
  There are 11 items in the scale. Each item is rated on a 5-point Likert scale from 0(not confident) to 4(a lot confident). The mean of 11 items multiplied by 25 represent the total score. The possible of the total score for the scale ranges from 0 [not confident] to 100 [extremely confident].
Decisional Conflict Scale | 1 hour after pre-test
  There are 16 items in the scale. Each item is rated on a 5-point Likert scale from 0(strongly agree) to 4(strongly disagree). The mean of 16 items multiplied by 25 represent the total score. The possible of the total score for the scale ranges from 0 [no decisional conflict] to 100 [extremely high decisional conflict]. Scores exceeding 37.5 are associated with decision delay.

CONTACTS AND LOCATIONS:
Overall Officials: Tsae Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen NH, Lin YP, Liang SY, Tung HH, Tsay SL, Wang TJ. Conflict when making decisions about dialysis modality. J Clin Nurs. 2018 Jan;27(1-2):e138-e146. doi: 10.1111/jocn.13890. Epub 2017 Jul 17. PMID 28543737
- [Background] Luque JS, Ross L, Gwede CK. Prostate Cancer Education in African American Barbershops: Baseline Client Survey Results and Differences in Decisional Conflict and Stage of Decision Making. Am J Mens Health. 2016 Nov;10(6):533-536. doi: 10.1177/1557988316630952. Epub 2016 Feb 9. PMID 26860126
- [Background] Catalona WJ, Richie JP, Ahmann FR, Hudson MA, Scardino PT, Flanigan RC, DeKernion JB, Ratliff TL, Kavoussi LR, Dalkin BL, Waters WB, MacFarlane MT, Southwick PC. Comparison of Digital Rectal Examination and Serum Prostate Specific Antigen in the Early Detection of Prostate Cancer: Results of a Multicenter Clinical Trial of 6,630 Men. J Urol. 2017 Feb;197(2S):S200-S207. doi: 10.1016/j.juro.2016.10.073. Epub 2016 Dec 22. PMID 28012755
- [Background] Groarke A, Curtis R, Walsh DMJ, Sullivan FJ. What predicts emotional response in men awaiting prostate biopsy? BMC Urol. 2018 Apr 24;18(1):27. doi: 10.1186/s12894-018-0340-9. PMID 29699543